CLINICAL TRIAL: NCT04767659
Title: Optical Monitoring of Neoadjuvant Chemotherapy and Prediction of Pathological Complete Response in Breast Cancer Patients
Brief Title: Monitoring Response to NAC and Prediction of pCR in Breast Cancer Patients Using Optical Imaging
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS San Raffaele (Other)
Collaborators: Politecnico di Milano (Other)
Responsible Party: Principal Investigator, Pietro Panizza, Head of Breast Imaging Unit, MD, IRCCS San Raffaele
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NADOPTIC
Record Dates: First submitted 2021-01-12; First posted 2021-02-23 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer Female; Chemotherapy Effect
Keywords: Neoadjuvant chemotherapy; Pathological complete response; Optical imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Women candidate for clinical trial (Experimental): Twenty adult women with a recent diagnosis of breast cancer, candidate for NAC, besides assessing the response to neoadjuvant chemotherapy using standard imaging evaluation, will undergo optical imaging at six selected time points from prior to commencement of NAC/baseline to the completion of NAC treatment (prior to surgery).
  Interventions: Device: MAMMOT2

INTERVENTIONS:
Device: MAMMOT2 — Breast cancer patients candidate for neoadjuvant chemotherapy will be evaluated with optical imaging prior to commencement of NAC/baseline, 2-5 days post-NAC, 6-8 days post-NAC, 2 weeks post-NAC, half-way through and on completion of NAC. 2 additional optical evaluations will be carried out on the first 5 patients enrolled, one before breast biopsy and one after the positioning of the metallic clip, in order to evaluate the potential artefacts related to these procedures.

SUMMARY:
Neoadjuvant chemotherapy (NAC) is the first line treatment for locally advanced breast cancer (BC). Besides making breast conserving surgery feasible, its main aim is to achieve a pathological complete response (pCR). Previous studies demonstrated that a pCR correlated with a higher disease-free survival. Tumor response may vary among different BC subtypes and only 30% of BC respond completely to NAC. Treating chemo-resistant disease with NAC may cause patient harm due to drug toxicity and surgery delay.

It is therefore very important to promptly identify those women who will not benefit from NAC.

Mammography and ultrasound proved ineffective in monitoring changes in lesion size due to therapy-induced fibrosis. MRI is the most accurate imaging technique for assessing early clinical response by measuring tumor size, however its accuracy is lower post NAC. This necessitates the need for a new technique able to non invasively assess the effectiveness of NAC. Optical techniques are sensitive to the biological changes that occur within the tumor after NAC administration. These changes occur prior to tumor size reduction.

Optically estimated total hemoglobin concentration correlates with the histological analysis of vasculature as well as with tumor-associated angiogenesis which can affect tumor changes during NAC. Other promising biomarkers related to tissue composition (water, lipid, collagen content) and structure (scattering) may also be evaluated by optical techniques.

The aim of the study is to monitor the effectiveness of NAC in BC patients with a near infrared spectroscopic imaging platform which allows to non-invasively detect changes in vascularization and size of BC and to characterize the presence of temporal changes in regional concentrations of relevant biomarkers (oxy- and deoxyhemoglobin, water, lipid and collagen concentration, scattering) within tissue during NAC.

This optical imaging technique will provide a non-invasive, safe and relatively inexpensive tool to monitor patients' response to NAC and to predict their outcome.

DETAILED DESCRIPTION:
In this study, an accurate, reliable, non-invasive modality with good patient tolerance will be tested to predict response to NAC in order to tailor the medical and surgical treatment.

The aim of this project is to monitor the effectiveness of NAC in BC patients with a new near infrared spectroscopic imaging platform which allows to non-invasively detect changes in size, vascularization and blood oxygenation in tumors and to characterize the presence of temporal changes in regional concentrations of relevant biomarkers like oxy- and deoxyhemoglobin, water, lipid and collagen and scattering in the tissue during NAC. This optical imaging tool will allow a non-invasive, safe and relatively inexpensive monitoring of NAC and prediction of patients' outcome.

A single-site, national, non-comparative, non-randomized study will be conducted at the San Raffaele Hospital in Milan in collaboration with the Politecnico di Milano. The medical device is a prototype developed by Politecnico di Milano.

Twenty adult women with a recent diagnosis of breast cancer and candidate for NAC, who fulfil the inclusion criteria and agree to voluntary participate in the study under informed consent, will be enrolled.

Besides assessing the response to neoadjuvant chemotherapy using conventional imaging evaluation (x-ray mammography and breast ultrasound prior to commencement/baseline, half way through and on completion of NAC; contrast-enhanced MRI prior to commencement/baseline and on completion of NAC), the patients enrolled will be evaluated with optical imaging at the following six selected time points (prior to commencement of NAC/baseline, 2-5 days post-NAC, 6-8 days post-NAC, 2 weeks post-NAC, half-way through and on completion of NAC).

A preliminary phase will be performed on the first 5 patients out of the 20 patients enrolled, in order to evaluate the potential artefacts related to a recent breast biopsy and to the positioning of a clip. In this preliminary phase, 2 additional optical evaluations will be carried out, one prior to the breast biopsy and one after the positioning of the clip.

Patients are enrolled in the study for the entire duration of NAC. No follow-up is required and patients will be followed according to the regular clinical standard of care. Moreover, the outcome of the optical investigation does not affect the treatment and management of the women enrolled in the study.

The duration of enrolment of the study is expected to be approximately 12 months. The study will end when the last patient enrolled will complete her chemotherapy treatment.

ELIGIBILITY:
Inclusion Criteria:

* Women above 18 years of age
* Women with a recent diagnosis of breast cancer candidate for neoadjuvant chemotherapy
* Women willing to give informed consent

Exclusion Criteria:

* Subject is pregnant or breastfeeding
* Subject is unable or unwilling to give informed consent
* Previous surgery of the same breast
* Presence of distant metastasis
* Breast implants

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-01-27 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Optical monitoring of neoadjuvant chemotherapy in breast cancer patients | The through completion study is that of an average of 1 year
  Optical data will be compared to the conventional imaging results and to the surgical specimen histology (gold standard)
Prediction of pathological complete response to neoadjuvant chemotherapy using optical imaging | The through completion study is that of an average of 1 year
  Optical data will be evaluated to distinguish responders from non responders

CONTACTS AND LOCATIONS:
Overall Officials: PANIZZA, Principal Investigator — IRCCS San Raffaele
Locations (1):
- Ospedale San Raffaele, Milan, Italy

REFERENCES:
- [Background] Wabnitz H, Taubert DR, Mazurenka M, Steinkellner O, Jelzow A, Macdonald R, Milej D, Sawosz P, Kacprzak M, Liebert A, Cooper R, Hebden J, Pifferi A, Farina A, Bargigia I, Contini D, Caffini M, Zucchelli L, Spinelli L, Cubeddu R, Torricelli A. Performance assessment of time-domain optical brain imagers, part 1: basic instrumental performance protocol. J Biomed Opt. 2014 Aug;19(8):086010. doi: 10.1117/1.JBO.19.8.086010. PMID 25121479
- [Background] Independent UK Panel on Breast Cancer Screening. The benefits and harms of breast cancer screening: an independent review. Lancet. 2012 Nov 17;380(9855):1778-86. doi: 10.1016/S0140-6736(12)61611-0. Epub 2012 Oct 30. PMID 23117178
- [Background] Brem RF, Lenihan MJ, Lieberman J, Torrente J. Screening breast ultrasound: past, present, and future. AJR Am J Roentgenol. 2015 Feb;204(2):234-40. doi: 10.2214/AJR.13.12072. PMID 25615743
- [Background] Liu B, Zheng Y, Huang G, Lin M, Shan Q, Lu Y, Tian W, Xie X. Breast Lesions: Quantitative Diagnosis Using Ultrasound Shear Wave Elastography-A Systematic Review and Meta--Analysis. Ultrasound Med Biol. 2016 Apr;42(4):835-47. doi: 10.1016/j.ultrasmedbio.2015.10.024. Epub 2016 Jan 6. PMID 26778289
- [Background] Durduran T, Choe R, Baker WB, Yodh AG. Diffuse Optics for Tissue Monitoring and Tomography. Rep Prog Phys. 2010 Jul;73(7):076701. doi: 10.1088/0034-4885/73/7/076701. PMID 26120204
- [Background] Leff DR, Warren OJ, Enfield LC, Gibson A, Athanasiou T, Patten DK, Hebden J, Yang GZ, Darzi A. Diffuse optical imaging of the healthy and diseased breast: a systematic review. Breast Cancer Res Treat. 2008 Mar;108(1):9-22. doi: 10.1007/s10549-007-9582-z. Epub 2007 Apr 28. PMID 17468951
- [Background] Taroni P, Pifferi A, Salvagnini E, Spinelli L, Torricelli A, Cubeddu R. Seven-wavelength time-resolved optical mammography extending beyond 1000 nm for breast collagen quantification. Opt Express. 2009 Aug 31;17(18):15932-46. doi: 10.1364/OE.17.015932. PMID 19724592
- [Background] Ferocino E, Martinenghi E, Dalla Mora A, Pifferi A, Cubeddu R, Taroni P. High throughput detection chain for time domain optical mammography. Biomed Opt Express. 2018 Jan 23;9(2):755-770. doi: 10.1364/BOE.9.000755. eCollection 2018 Feb 1. PMID 29552410
- [Background] Quarto G, Spinelli L, Pifferi A, Torricelli A, Cubeddu R, Abbate F, Balestreri N, Menna S, Cassano E, Taroni P. Estimate of tissue composition in malignant and benign breast lesions by time-domain optical mammography. Biomed Opt Express. 2014 Sep 18;5(10):3684-98. doi: 10.1364/BOE.5.003684. eCollection 2014 Oct 1. PMID 25360382
- [Background] Taroni P, Quarto G, Pifferi A, Ieva F, Paganoni AM, Abbate F, Balestreri N, Menna S, Cassano E, Cubeddu R. Optical identification of subjects at high risk for developing breast cancer. J Biomed Opt. 2013 Jun;18(6):060507. doi: 10.1117/1.JBO.18.6.060507. PMID 23804215
- [Background] Taroni P, Paganoni AM, Ieva F, Pifferi A, Quarto G, Abbate F, Cassano E, Cubeddu R. Non-invasive optical estimate of tissue composition to differentiate malignant from benign breast lesions: A pilot study. Sci Rep. 2017 Jan 16;7:40683. doi: 10.1038/srep40683. PMID 28091596
- [Background] Pearlman PC, Adams A, Elias SG, Mali WP, Viergever MA, Pluim JP. Mono- and multimodal registration of optical breast images. J Biomed Opt. 2012 Aug;17(8):080901-1. doi: 10.1117/1.JBO.17.8.080901. PMID 23224161
- [Background] Tavakoli B, Zhu Q. Two-step reconstruction method using global optimization and conjugate gradient for ultrasound-guided diffuse optical tomography. J Biomed Opt. 2013 Jan;18(1):16006. doi: 10.1117/1.JBO.18.1.016006. PMID 23296038